CLINICAL TRIAL: NCT02082821
Title: Pure-Heart-1: A P2X7R Single Nucleotide Mutation Promotes Chronic Allograft Vasculopathy
Brief Title: A P2X7R Single Nucleotide Mutation Promotes Chronic Allograft Vasculopathy
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Paolo Fiorina, Assistant Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: Pure-Heart-1; 14GRNT1873002 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2014-03-05; First posted 2014-03-10 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Cardiac Allograft Vasculopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood mononulcear cells
Oversight: Data Monitoring Committee: No

SUMMARY:
Heart transplantation (HT) is a lifesaving procedure for patients with end-stage heart failure and provides a better survival and quality of life if compared to medical treatment. HT is subject to alloimmune response, which, if left uncontrolled, is capable of jeopardizing long-term cardiac function. Advances in immunosuppression have enhanced the survival of HT patients. Nearly 2500 HT per year have been performed in the US during the last 10 years and despite significant improvements, long-term survival rates remain poor. More than 20% of patients do not survive more than 3 years, and those who survive are afflicted by long-term complications of alloimmunity and chronic immunosuppression. Life expectancy of patients who lose cardiac allografts is dramatically poor due to the absence of any therapeutic tool apart from re-transplantation, which is plagued by poor outcomes. The identification of novel therapeutic targets is thus mandatory. ATP/P2X7R signaling in T cells is highly relevant for cardiac allograft survival. ATP is a small molecule present at high concentrations inside cells; it is released as extracellular ATP (eATP) following cell damage or death where it acts as a danger signal. ATP is sensed by the P2X receptors (seven receptors named P2X1-7), mainly expressed by T lymphocytes. We have recently demonstrated that the ATP/P2X7R axis has a key role in cardiac allograft survival in humans and mice. Cardiac allograft vasculopathy (CAV) is a major limiting factor for HT survival; indeed CAV occurs in 50% of HT recipients by 5 years after transplantation and invariably results in allograft failure. CAV is clearly of immunological origin, as syngeneic murine grafts do not develop it. Once CAV occurs, the most definitive treatment is re-transplantation, but survival remains poor. We hypothesize that a single nucleotide polymorphysm (SNP) loss-of-function P2X7R mutation (p.Glu496Ala / c.1513A>C, rs3751143) generates a compensatory upregulation of the other purinergic receptors (P2XsR), thus creating a state of hypersensitivity to eATP. This eATP hypersensitivity results in an abnormal generation of Th1/Th17 cells, that leads to CAV and early cardiac allograft loss. Our study will answer a fundamental question: What is the effect of the P2X7R loss-of-function mutation on the immune system? Our goal is to generate the first targeted-therapy for a selected group of cardiac transplant recipients.

DETAILED DESCRIPTION:
Heart transplantation is a lifesaving procedure however, more then 20% of patients do not survive beyond 3 years, being the cardiac allograft afflicted by cardiac allograft vasculopathy (CAV), which results in allograft loss. The purine adenosine 5'-triphosphate (ATP), released during cell damage/inflammation, is sensed by the ionotropic purinergic P2X7 receptor (P2X7R), which is expressed primarily, though not exclusively, on lymphocytes, thus regulating T cell activation. Loss-of-function single nucleotide mutations (SNPs) have been detected for P2X7R gene; particularly the Glu496 to Ala 1513A>C (rs3751143) P2X7R loss-of-function mutation is relatively common (1-3% of individuals are mutated omozygous and 25% are heterozygous). Our central hypothesis is that a loss-of-function P2X7R mutation identifies a group of cardiac transplanted patients at high risk for CAV and cardiac allograft loss because of a compensatory overexpression of P2X1R/P2X4R, which induces a disregulation of T-bet/ROR-g, ultimately leading to the abnormal generation of Th1/Th17 cells. Our primary goal is to define the effect of the P2X7R loss-of-function mutation on clinical end points in the CTOT-05 cohort of cardiac transplant recipients (200 patients) and to explore the effects of the mutation on the immune system. Our preliminary data demonstrated that P2X7R increases during cardiac transplant rejection in vivo in mice and in humans and it is activated by ATP released by cardiac cells, thus triggering activation of Th1/Th17 cells. However, while short-term disruption of the P2X7R pathway prolongs cardiac allograft survival, the genetic deletion of P2X7R accelerates CAV and shortens cardiac allograft survival. This was evident in P2X7R KO-B6 mice and in a group of cardiac transplant recipients bearing the P2X7R loss-of-function mutation. Based on our published results and our novel observations, we have developed the following working hypothesis: P2X7R loss-of-function mutation generates a compensatory overexpression of the other ionotropic purinergic receptors (P2X1/P2X4) with chronic delivery of ATP immunity, hyperactivation T-bet/ROR-g, abnormal generation of Th1/Th17 cells and ultimately leading to accelerated CAV and to cardiac allograft loss. To test this hypothesis, we will follow two main paths: i) we will evaluate in the CTOT-05 cohort of cardiac transplant recipients the effect of the Glu496 to Ala 1513A>C (rs3751143) P2X7R loss-of-function mutation on clinical end points (development of coronary artery vasculopathy, death, re-transplantation or re-listed for transplantation, any rejection) in the first year post transplant; ii) we will explore in vivo and ex vivo in the CTOT-05 cohort of cardiac transplant recipients the effects of P2X7R loss-of-function mutation on the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Male or female cardiac recipients
* 18-65 years of age
* undergoing primary heart transplantation
* the graft must be functional at the time of randomization.
* patient willing and capable of giving written informed consent for study participation and anticipated to be able to participate in the study for 12 months

Exclusion Criteria:

* Recipient of multi-organ transplants or previously transplanted organs
* Patients with donor greater than 65 years
* Donor heart cold ischemic time > 6 hours.
* Patients who are recipients of ABO incompatible transplants
* Patients with platelet count < 50,000/mm3 at the evaluation before transplantation
* Patient who have received an unlicensed drug or therapy within one month prior to study entry or if such therapy is to be instituted post-transplantation
* Patient with a current severe systemic infection
* Patient unable to participate in the study for the full 12-month period
* Presence of severe hypercholesterolemia (≥ 350 mg/dL; ≥ 9 mmol/L) or hypertriglyceridemia (≥ 750 mg/dL; ≥ 8.5 mmol/L)
* Patients with any past (within the past 5 years) or present malignancy (other than excised basal cell carcinoma)
* Females capable of becoming pregnant must have a negative pregnancy test prior to randomization and are required to practice a medically approved method of birth control for the duration of the study and a period of 8 weeks following discontinuation of study medication, even where there has been a history of infertility.
* Patients with HIV, hepatitis B or C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the CTOT-05 cohort of cardiac transplant recipients will be stratified according to the genotype (P2X7R+/+, P2X7R+/- and P2X7R-/-) and compared for the development of CAV
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-01; Primary Completion 2019-08 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Cardiac Allograft Vasculopathy | 1 year
  nominal change from baseline to 1 year in percent atheroma volume measured by intravascular ultrasound

SECONDARY OUTCOMES:
Heart Rejection or Patient Death | 6 months; 12 months
  * Death
  * re-transplant
  * biopsy proven acute rejection
  * antibody mediated rejection
  * cellular rejection;
  * treated rejection
  * hemodynamic compromise-associated rejection
  * chronic allograft vasculaopathy at 12-months
  * total atheroma volume; change in average maximal intimal thickness
  * rapid progressive chronic allograft vasculaopathy (change in maximal intimal thickness) ≥0.5 mm in the first year (intravascular ultrasound)
  * histological changes of antibody mediated rejection (Immunohistochemistry).

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Fiorina, MD PhD, Principal Investigator — Boston Children's Hospital, Harvard Medical School
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No